CLINICAL TRIAL: NCT05774392
Title: An Observational Study of Patients With Chronic Kidney Disease
Status: Withdrawn | Type: Observational
Why Stopped: This protocol never enrolled any paticipants
Sponsor: Target PharmaSolutions, Inc. (Industry)
Responsible Party: Sponsor
Other Study IDs: TARGET-KIDNEY
Record Dates: First submitted 2023-03-07; First posted 2023-03-17 (Actual); Last update posted 2025-12-17 (Actual); Status verified 2025-12

CONDITIONS: Kidney Disease, Chronic; End Stage Kidney Disease
MeSH Terms: conditions — Renal Insufficiency, Chronic; Kidney Failure, Chronic | interventions — Watchful Waiting

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Other
Biospecimen Retention: Samples With DNA — Whole blood serum
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Disease Cohort
  Interventions: Other: Observational
- Engaged Cohort
  Interventions: Other: Observational

INTERVENTIONS:
Other: Observational — Observational

SUMMARY:
TARGET-KIDNEY is an observational research study to conduct a comprehensive review of outcomes for patients with chronic kidney disease (CKD) and end-stage renal disease (ESKD).

ELIGIBILITY:
Disease Cohort

Inclusion Criteria:

* Adult* patients at the time of enrollment with a diagnosis of CKD/ESKD by ICD-10 code in the EHR interface

Exclusion Criteria:

* Death
* Manual removal (sponsor or site request)
* No EHR interface encounter > 3 years

Engaged Cohort

Inclusion Criteria:

* Adult * patients diagnosed and managed for CKD/ESKD invited to participate
* Ability to provide written informed consent

Exclusion Criteria:

* Patient expressed desire to withdraw consent to complete PROs
* Failure to complete PROs within 24 weeks of initial invitation
* Greater than 24 months lapse of survey completion after baseline surveys completed
* Additionally, the criteria detailed for Disease Cohort apply to the Engaged Cohort

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: The study will include adults who are being managed for Stage 1-5 CKD or received a transplant for ESKD.
Sampling Method: Non-Probability Sample
Enrollment: 0 (Actual)
Dates: Start 2025-04 (Estimated); Primary Completion 2025-04-07 (Actual); Study Completion 2025-04-07 (Actual)

PRIMARY OUTCOMES:
To characterize the natural history of disease in patients with CKD/ESKD. | 20 Years
To assess safety and effectiveness of CKD/ESKD treatments and treatments for complications of either condition | 20 Years

SECONDARY OUTCOMES:
To evaluate provider management practices in the treatment of patients with CKD/ESKD | 20 Years
To evaluate longitudinal and patient reported outcomes in CKD/ESKD | 20 Years
To select and evaluate quality of care measures for patients with CKD/ESKD | 20 Years

IPD SHARING:
Plan to Share IPD: Undecided